CLINICAL TRIAL: NCT06174597
Title: Efficacy and Safety of Umbilical Cord Artery-derived Perivascular Stem Cells in Patients With Critical Limb Ischemia
Brief Title: Umbilical Cord Artery-derived Perivascular Stem Cells for the Critical Limb Ischemia Therapy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nanjing University (Other)
Responsible Party: Principal Investigator, Li-jun Ding, principal investigator, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CLI-2023
Record Dates: First submitted 2023-07-19; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-07

CONDITIONS: Critical Limb Ischemia
Keywords: Critical Limb Ischemia; Umbilical cord artery-derived perivascular stem cells
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UCA-PSCs/bFGF group (Experimental): Clusters of umbilical cord artery-derived perivascular stem cells (Dose: 1.2 x 10^8 cells+20ng bFGF /20mL/vial)
  Interventions: Procedure: UCA-PSCs/bFGF or bFGF Intramuscular injection
- bFGF group (Active Comparator): (Dose: 20ng bFGF /20 mL/vial)
  Interventions: Procedure: UCA-PSCs/bFGF or bFGF Intramuscular injection

INTERVENTIONS:
Procedure: UCA-PSCs/bFGF or bFGF Intramuscular injection — After skin disinfection, according to the distribution characteristics of blood vessels around the vascular lesion area, the site that is most likely to establish a new collateral circulation in vascular anatomy is selected. According to the vascular lesion of each subject, 40 reasonable injection sites are selected for Clusters of umbilical cord artery-derived perivascular stem cells with bFGF or bFGF only.

SUMMARY:
This clinical trial included 2 periods. During the first period, it was a single arm study to explore the safety of umbilical cord artery-derived stem cells (UCA-PSCs) in the treatment of patients with critical limb ischemia (CLI). During the second perid, it was a single-center, randomized, controlled prospective study to determine the efficacy of the UCA-PSCs treatment. Those who had CLI were enrolled in the study.

DETAILED DESCRIPTION:
According to the enrollment and exclusion criteria, the patients were enrolled.During the first period, 10 patients were injected with UCA-PSCs/bFGF, a second injection was given 8 weeks later. During the second period, the patients were randomly divided into two groups by computer randomization.Group A was the UCA-PSCs/bFGF group (test group). Group B was the bFGF group (control group).

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 80, of any gender;
2. Diagnosed with lower extremities ischemia, classified as Rutherford Stage IV-V, affecting at least one limb. If both lower limbs have ischemic disease, the researcher will determine which affected limb will be studied. The resting ankle systolic pressure (dorsalis pedis artery or posterior tibial artery) of the affected limb is less than 60mmHg, or the toe systolic pressure is less than 40 mmHg, or the Ankle-Brachial Index (ABI) is less than 0.50;
3. Within the last month, Digital Subtraction Angiography (DSA), Computed Tomography Arteriography (CTA), Magnetic Resonance Angiography (MRA)，or vascular ultrasound has confirmed that one or more of the arteries (superficial femoral artery, i.e., the femoral artery below the deep femoral artery branch, the popliteal artery, and its following arteries) have a stenosis of ≥75% or occlusion;
4. Patient experiences rest pain in the limb due to ischemia for at least two weeks;
5. Inoperable or not suitable for endovascular treatment，or no obvious improvement after surgical treatment;
6. Expected lifespan >2 years;
7. Good compliance, accepting dietary control and medication treatment, with an informed consent form signed by the patient themselves or their legal representatives.

Exclusion Criteria:

1. Acute ischemic disease of the lower limb(s) occurred within the past 2 weeks, or patients with acute progression of lower extremity arterial ischemic disease, or those with local/diffuse gangrene;
2. Unsatisfactory evaluation of condition stability after vascular reconstruction surgery or sympathetic nerve removal surgery performed within 4 weeks，or possibility of undergoing amputation in the next 4 weeks;
3. Stenosis of ≥75% in the main-iliac artery;
4. Diabetic patients with HbA1c > 10%;
5. Abnormal laboratory test results that meet any of the following criteria:i. Abnormal blood routine examination: Hemoglobin (HGB)<80 g/L, or white blood cell count (WBC)<3.0×10^9/L, or platelet count (PLT)<50×10^9/L; ii. Abnormal liver function: Aspartate aminotransferase (AST)>2 times the upper limit of normal (ULN), or alanine aminotransferase (ALT)>2×ULN, total bilirubin (TBIL)>2×ULN; iii. Severe renal dysfunction requiring dialysis treatment;iv. Other abnormal laboratory testing indicators that researchers believe may affect the evaluation of trial results;
6. Diseases unsuitable for clinical trials, or contraindications to surgery: i. Difficult-to-control hypertension (>180/110mmHg), severe heart failure (NYHA IV), or EF<30%;ii. Patients who have had a stroke, brain hemorrhage, myocardial infarction, or unstable angina in the past one month; iii. Patients with malignant tumors;iv. Receiving immunosuppressants, hemodialysis, chemotherapy, and radiotherapy; v. Active infection, HIV antibody positive, Hepatitis C antibody positive, Hepatitis B (HBsAg positive and Hepatitis B virus DNA quantitative detection value greater than 1×10^3 IU/mL); vi. Serious infections (like cellulitis, osteomyelitis etc.) in the observational limb, exposure of distal fascia or skeleton, unable to maintain wound care for ulcers in the surgical area etc.; vii. History of major surgery or serious injury within the last one months;
7. During the trial, taking the following drugs at doses greater than stated below, except those who stop medication or adjust the dose to the prescribed dose for 7 days according to the washout period: i. COX-2 inhibitor drugs (such as nimesulide); ii. Aspirin (more than 100 mg/day);iii. High-dose steroid medications, excluding inhaled steroids; iv. Opioid analgesics (like morphine) for 2 weeks or longer;
8. Congenital or acquired immunodeficiency;
9. Pregnant women or those planning pregnancy;
10. Diseases like pulmonary heart disease and mental illness that researchers believe are unstable and cannot complete the trial, or comorbidities that could interfere with safety checks and effectiveness assessments;
11. Currently participating in other clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
hindlimb flow index | 24 months
  measured by Laser Doppler

SECONDARY OUTCOMES:
Increase in transcutaneous partial oxygen pressure (TcPO2) | 24 months
  measured by Doppler
Ankle brachial pressure index (ABPI) | 24 months
  measured by Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Haiming Xia, phD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- The affiliated Drum Towel Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China